CLINICAL TRIAL: NCT06523049
Title: A Prospective, Multicenter, Phase II Clinical Trial of Vorolanib in Combination With Sintilimab for Advanced Renal Cell Carcinoma After Failure of Prior Immune Checkpoint Inhibitors Based Combination Therapy
Brief Title: Vorolanib Plus Sintilimab for Advanced Renal Cell Carcinoma After Failure of Prior Immune Checkpoint Inhibitors Based Combination Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hao Zeng (Other)
Responsible Party: Sponsor-Investigator, Hao Zeng, Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VORSIN-RCC
Record Dates: First submitted 2024-07-14; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Renal Cell Carcinoma; Immunotherapy; Molecular Targeted Therapy
Keywords: Vorolanib; Sintilimab
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — vorolanib; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination treatment group (Experimental): Participants in this group will receive vorolanib tablets, 200 mg orally once daily, plus sintilimab injection, 200 mg intravenously every three weeks.
  Interventions: Drug: Vorolanib Tablets; Drug: Sintilimab Injection

INTERVENTIONS:
Drug: Vorolanib Tablets — Multi-targeted receptor tyrosine kinase inhibitor with potent inhibition of VEGFR2, KIT, PDGFR, FLT3 and RET, exerting anti-tumor effects mainly through inhibition of neovascularization.
  Other Names: Vorolanib
Drug: Sintilimab Injection — Recombinant human-derived immunoglobulin G (IgG4)-type anti-programmed cell death receptor-1 (PD-1) monoclonal antibody, by binding to PD-1 and blocking PD-1 binding to PD-L1 and PD-L2, disarms the immunosuppressive effect, activates T-cell function, and enhances T-cell immunosurveillance and killing ability against tumors to generate tumor immune response.
  Other Names: Sintilimab

SUMMARY:
This Phase II trial assesses Vorolanib and Sintilimab for advanced renal cell carcinoma after previous therapy failure. Participants receive the treatment until disease progression, intolerable side effects, death, or withdrawal. The primary endpoint is progression-free survival (PFS).

DETAILED DESCRIPTION:
This is a Phase II, multicenter, single-arm clinical trial designed to assess the efficacy and safety of Vorolanib in combination with Sintilimab in treating advanced renal cell carcinoma following the failure of prior immune checkpoint inhibitors based combination therapy. Participants will continue to receive Vorolanib and Sintilimab until disease progression, development of unacceptable toxic effects, death, or if the physician or patient decides to withdraw from the study. The primary endpoint is progression-free survival (PFS) according to RECIST v1.1 criteria as evaluated by the investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤75 years, any gender.
2. Histologically confirmed diagnosis of renal cell carcinoma.
3. Diagnosis of metastatic renal cell carcinoma or TNM stage IV (according to the 2017 TNM staging system). Evidence of distant metastasis by imaging or pathology.
4. Prior immune checkpoint inhibitors based combination therapy, dual immune combination, or immune monotherapy with disease progression, or who have received second/third line targeted monotherapy, immune monotherapy, or a change in immune-based combination therapy after failure of one of the above therapies for no more than 1 month and have completed the washout period. ECOG performance status ≤2.
5. Life expectancy of at least 3 months.
6. Signed informed consent and ability to comply with the protocol-specified visits and procedures.
7. Agreement to provide tumor tissue and blood specimens required for the study.
8. Adequate organ and bone marrow function as follows: absolute neutrophil count (ANC) ≥1×10^9/L, platelets (PLT) ≥50×10^9/L, hemoglobin (HGB) ≥80g/L; liver function: serum total bilirubin (TBIL) ≤3 times the upper limit of normal (ULN), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤5 times ULN, serum albumin (ALB) ≥20 g/L; renal function: serum creatinine (Cr) ≤3×ULN.

Exclusion Criteria:

1. Pathologically diagnosed with non-renal cell carcinoma, collecting duct carcinoma.
2. First-line treatment with targeted monotherapy, or progression after first-line immune checkpoint inhibitors based combination therapy, followed by more than 1 month of treatment with targeted therapies, anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-PD-L2 antibodies, or anti-CTLA-4 antibodies specifically targeting T cell co-stimulation or checkpoint pathways and/or incomplete washout period.
3. Active brain metastases.
4. Personal history of other malignant tumors within 3 years with a different primary site or histology than that being evaluated in this study, excluding patients with well-controlled basal cell carcinoma, squamous cell carcinoma, or cervical intraepithelial neoplasia.
5. Major surgery or severe trauma within 4 weeks prior to enrollment.
6. Subjects with conditions requiring systemic corticosteroids (>10mg/day prednisone or equivalent) or other immunosuppressive medications within 14 days prior to initial study drug administration. Subjects with inactive autoimmune disease are allowed to receive local, ophthalmic, intra-articular, intranasal, inhaled corticosteroids, or adrenal replacement steroids (>10mg/day prednisone dose or equivalent).
7. Known or suspected active autoimmune disease (congenital or acquired), such as interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, thyroiditis, etc. Subjects with type 1 diabetes, thyroid dysfunction requiring only hormone replacement therapy, skin diseases (such as vitiligo, psoriasis, or alopecia) that do not require systemic treatment, or conditions expected not to recur in the absence of external triggering factors are allowed to participate in this study. Known allogeneic organ transplant (excluding corneal transplant) or allogeneic hematopoietic stem cell transplant.
8. Allergy to any component of monoclonal antibodies.
9. Uncontrolled other severe diseases, including but not limited to:

   1. Severe infection in the active or poorly controlled clinical phase;
   2. HIV infection (HIV antibody positive);
   3. Acute or chronic active hepatitis B (HBsAg positive and HBV DNA >1*103/ml) or acute or chronic active hepatitis C (HCV antibody positive and HCV RNA >15IU/ml);
   4. Active pulmonary tuberculosis, etc.
10. NYHA class III-IV congestive heart failure, persistent symptomatic arrhythmia, uncontrolled atrial fibrillation; multiple echocardiographic assessments of left ventricular ejection fraction (LVEF) lower than the lower limit of normal.
11. Uncontrolled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg);
12. Any arterial thrombosis, embolism, or ischemia in the past 6 months prior to enrollment, such as myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, etc.;
13. Diseases requiring warfarin (coumarin) anticoagulant therapy;
14. Uncontrolled hypercalcemia (calcium ion >1.5 mmol/L or calcium >12 mg/dL or corrected serum calcium >ULN), or symptomatic hypercalcemia requiring continued bisphosphonate therapy;
15. Uncontrolled adrenal insufficiency;
16. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months;
17. Severe, non-healing wounds or ulcers;
18. Gastrointestinal diseases with impaired gastrointestinal function (such as malabsorption, ulcerative disease, uncontrollable nausea, vomiting, diarrhea, or small bowel resection);
19. Other acute or chronic diseases, mental illnesses, or laboratory abnormalities that may lead to the following outcomes: increased risk associated with study participation or drug administration, or interference with interpretation of study results, and deemed ineligible for study participation at the discretion of the investigator;
20. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 3 years
  Progression-free survival is assessed by investigators based on RECIST1.1, including disease progression or death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 3 years
  Objective response rate is the proportion of participates with complete response (CR) or partial response (PR), based on RECIST1.1.
Overall Survival (OS) | 3 years
  Overall survival is the time from starting treatment to still being alive.
Adverse Events (AEs) | 3 years
  Adverse events are the incidence of treatment-emergent adverse events as assessed by CTCAE v5.0, including type and severity.
Disease Control Rate (DCR) | 3 years
  Disease control rate is the proportion of participates with complete response (CR), partial response (PR) or stable disease (SD), based on RECIST1.1.
Duration of Response (DoR) | 3 years
  Duration of response is the time from first response (complete or partial response) to disease progression or death.
Quality of Life (QoL) assessed by FKSI-19 | 3 years
  Quality of life is assessed by FKSI-19
Quality of Life (QoL) assessed by EQ-5D-5L | 3 years
  Quality of life is assessed by EQ-5D-5L.
Pain Score | 3 years
  Evaluate pain using visual analogue scale (VAS), range from 0 to 10, higher scores predict a poor prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Zeng, Doctor, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data would be available starting from the time when summary data are published or otherwise made available, for 3 years.
Access Criteria: Other researchers access the data by sending an email to our PI.

REFERENCES:
- [Background] Ljungberg B, Albiges L, Abu-Ghanem Y, Bedke J, Capitanio U, Dabestani S, Fernandez-Pello S, Giles RH, Hofmann F, Hora M, Klatte T, Kuusk T, Lam TB, Marconi L, Powles T, Tahbaz R, Volpe A, Bex A. European Association of Urology Guidelines on Renal Cell Carcinoma: The 2022 Update. Eur Urol. 2022 Oct;82(4):399-410. doi: 10.1016/j.eururo.2022.03.006. Epub 2022 Mar 26. PMID 35346519
- [Background] Liang C, Yuan X, Shen Z, Wang Y, Ding L. Vorolanib, a novel tyrosine receptor kinase receptor inhibitor with potent preclinical anti-angiogenic and anti-tumor activity. Mol Ther Oncolytics. 2022 Jan 10;24:577-584. doi: 10.1016/j.omto.2022.01.001. eCollection 2022 Mar 17. PMID 35252556
- [Background] Pei Dong et al. , Anlotinib combined with sintilimab as first-line treatment in patients with advanced non-clear cell renal cell carcinoma (nccRR): Preliminary results from an exploratory prospective multicentre clinical study.. JCO 42, 4544-4544(2024). DOI:10.1200/JCO.2024.42.16_suppl.4544
- [Background] Lee CH, Shah AY, Rasco D, Rao A, Taylor MH, Di Simone C, Hsieh JJ, Pinto A, Shaffer DR, Girones Sarrio R, Cohn AL, Vogelzang NJ, Bilen MA, Gunnestad Ribe S, Goksel M, Tennoe OK, Richards D, Sweis RF, Courtright J, Heinrich D, Jain S, Wu J, Schmidt EV, Perini RF, Kubiak P, Okpara CE, Smith AD, Motzer RJ. Lenvatinib plus pembrolizumab in patients with either treatment-naive or previously treated metastatic renal cell carcinoma (Study 111/KEYNOTE-146): a phase 1b/2 study. Lancet Oncol. 2021 Jul;22(7):946-958. doi: 10.1016/S1470-2045(21)00241-2. Epub 2021 Jun 15. PMID 34143969
- [Background] Laccetti AL, Garmezy B, Xiao L, Economides M, Venkatesan A, Gao J, Jonasch E, Corn P, Zurita-Saavedra A, Brown LC, Kao C, Kinsey EN, Gupta RT, Harrison MR, Armstrong AJ, George DJ, Tannir N, Msaouel P, Shah A, Zhang T, Campbell MT. Combination antiangiogenic tyrosine kinase inhibition and anti-PD1 immunotherapy in metastatic renal cell carcinoma: A retrospective analysis of safety, tolerance, and clinical outcomes. Cancer Med. 2021 Apr;10(7):2341-2349. doi: 10.1002/cam4.3812. Epub 2021 Mar 1. PMID 33650321
- [Background] Iacovelli R, Ciccarese C, Procopio G, Astore S, Cannella MA, Maratta MG, Rizzo M, Verzoni E, Porta C, Tortora G. Current evidence for second-line treatment in metastatic renal cell carcinoma after progression to immune-based combinations. Cancer Treat Rev. 2022 Apr;105:102379. doi: 10.1016/j.ctrv.2022.102379. Epub 2022 Mar 12. PMID 35303548
- See also: A Trial of Lenvatinib (E7080) Plus Pembrolizumab in Participants With Selected Solid Tumors (NCT02501096) — http://clinicaltrials.gov/study/NCT02501096?term=NCT02501096&rank=1